CLINICAL TRIAL: NCT04195789
Title: Assessment of Interstitial Lung Disease in Rheumatoid Arthritis by Lung Ultrasound
Acronym: PO-PID
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0859
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Lung Diseases; Lung Diseases, Interstitial; Rheumatoid Arthritis
MeSH Terms: conditions — Lung Diseases; Lung Diseases, Interstitial; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * In routine care a blood test (blood count, platelets, ionogram, VS (velocity sedimentation), CRP (C reactive protein), liver test, BNP (B-type natriuretic peptide), electrophoresis of serum proteins, quantiferon, HIV serologies, HBV : hepatitis B virus , HCV: hepatitis C virus) will be performed on the day of inclusion visit (V0).
  * Two more tubes of 4cc will be collected for a serum bank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sample population: Patients with Rheumatoid Arthritis consultant for the start of a biotherapy or targeted therapy agreeing to participate.
  Interventions: Other: Lung sonography

INTERVENTIONS:
Other: Lung sonography — Realization of a lung sonography with scoring of the number of B-lines exploring 14 intercostal spaces.
  Duration of the exam : twenty minutes. Recording for a second analysis by another lung specialist.

SUMMARY:
The high resolution chest scan is the gold standard for the screening of interstitial lung disease, but this remains an onerous examination, and irradiating.

Ultrasound could be used to detect these disorders with a very good sensitivity and specificity. This exam offers the advantage of being non radiating, inexpensive, and accessible to the rheumatologist who already uses it in their daily practice.

The investigators want to assess the lung ultrasound performance compared with the gold standard.

Patients will be included during a regular follow-up consultation with their referent rheumatologist. If there is an indication of first line biotherapy or targeted therapy the doctor will propose to the patient to participate in the study, give him the information leaflet, collect orally non-opposition, and will complete a survey for evaluation of the general health and potential risk factors for interstitial lung.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18
* With rheumatoid arthritis meeting the criteria ACR (American College of Rheumatology)/ EULAR (EUropean League Against Rheumatism) 2010
* Never received any biotherapy or targeted therapy
* Having an indication of introduction of biotherapy or therapy targeted (JAK inhibitors) (JAK : Janus kinase)

Exclusion Criteria:

* Refusal to participate in the study
* Known pulmonary disease that can alter lung interstitium: cardiac decompensation, COPD (chronic obstructive pulmonary disease), thoracic surgery, infection pulmonary
* Patient with respiratory functional signs suggestive of PID (Diffuse interstitial lung disease)
* Patient with signs of cardiac decompensation
* Patient with pulmonary auscultation suggestive of PID
* Pregnant or lactating woman
* Psychiatric pathology seriously hindering understanding
* Difficulty understanding oral French
* Person deprived of liberty or under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for a rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Sensibility and specificity of the lung sonography for interstitial lung disease screening in rheumatoid arthritis patients. | Month 12
  To estimate the sensitivity and specificity of pulmonary ultrasound compared to CT scans in patients with rheumatoid arthritis consulting at the Lyon South Hospital Centre or the Edouard Herriot Hospital for the start-up of biotherapy or targeted therapy. (CT : computerized tomography)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Rhumatologie. Centre hospitalier Lyon Sud. 69310, Pierre-Bénite, France